CLINICAL TRIAL: NCT04915625
Title: A Prediction Model of 28-day Mortality in Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0603
Record Dates: First submitted 2021-06-04; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Septic Shock
Keywords: mortality; Predictive model
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Death group: Retrospective observational studies
- Survival group: Retrospective observational studies

SUMMARY:
This clinical study adopts the design of cohort research, selects the sepsis shock patients admitted to our hospital ICU as the research object, takes the 28-day mortality rate as the outcome index, collects the baseline data of the patient, the severity of the disease, vital signs, the main infection site, the laboratory-related index, the treatment method and other data, screens out the risk factors affecting the sepsis shock 28-day mortality rate and constructs the prediction model accordingly, analyzes the prediction model with the subject's working characteristic curve (ROC). The recognition ability of the model is calculated by the area under the ROC curve (AUC) and the ability of the model to predict 28-day mortality with SOFA and APACHE II.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age, gender-neutral;
2. Diagnosed with sepsis shock;
3. ICU survives longer than 48 h;
4. The preservation of clinical data is complete;

Exclusion Criteria:

- Diagnosed with sepsis shock within 6 hours of emergency treatment; Combined with people with autoimmune diseases; 3. Organ transplantation or immunosuppressive treatment; 4. Severe heart, liver and kidney insufficiency; 5. Late stage of malignant tumor; 6. Maternity; 7. Referral or referral to another hospital;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sepsis shock patients admitted to our hospital
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
All causes of 28 days mortality | 28 days
  The all-cause mortality rate is measured from the time the ICU is admitted to the hospital and 28 days after admission (regardless of ICU, hospitalization or out-of-hospital mortality).

SECONDARY OUTCOMES:
ICU hospitalization time | 2 years
  hospitalization time
hospitalization mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: ZHIJUN XU, MS, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No